CLINICAL TRIAL: NCT06451055
Title: Effect of Dietary Energy Restriction on Reversing Isolated Impaired Fasting Glucose: A Proof of Concept Study
Brief Title: Low-calorie Diet in Isolated Impaired Fasting Glucose
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sathish Thirunavukkarasu, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00007848
Record Dates: First submitted 2024-05-31; First posted 2024-06-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Isolated Impaired Fasting Glucose
Keywords: Low-calorie diet; Prediabetes; Overweight; Obesity; Fasting hyperglycemia
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Nursing staff conducting outcome assessments and laboratory personnel will be blinded to participants' treatment status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-calorie diet (Experimental): Participants following a low-calorie diet (LCD) consisting of approximately 1,300 kcal/day (37% carbohydrates, 25% protein, 39% fat, and 7 g of fiber per meal) over an eight-week period.
  Interventions: Behavioral: Low-calorie diet
- Routine dietary and physical activity habits (Active Comparator): Control participants are asked to maintain their routine dietary and physical activity habits.
  Interventions: Behavioral: Routine dietary and physical activity habits

INTERVENTIONS:
Behavioral: Low-calorie diet — The low-calorie diet consists of approximately 1,300 kcal/day (37% carbohydrates, 25% protein, 39% fat, and 7 g of fiber per meal) over an eight-week period. Participants receive weekly pre-prepared meals from Trifecta Nutrition (Trifecta Inc. California, USA) with options for breakfast, lunch, and dinner, meticulously crafted by certified dieticians and expert chefs. Participants are encouraged to consume 1-2 liters of water daily and maintain their habitual physical activity levels.
  Other Names: Dietary energy restriction
  Arms: Low-calorie diet
Behavioral: Routine dietary and physical activity habits — Participants are asked to maintain their habitual dietary and physical activity habits for the 8-week study period.
  Arms: Routine dietary and physical activity habits

SUMMARY:
This study aims to evaluate the preliminary efficacy of a low-calorie diet (LCD) intervention in addressing the underlying pathophysiological abnormalities and improving fasting hyperglycemia among individuals with isolated impaired fasting glucose (i-IFG). Additionally, it seeks to assess the feasibility and acceptability of the LCD intervention.

DETAILED DESCRIPTION:
This proof-of-concept randomized controlled trial (RCT) will enroll 34 individuals aged 35-65 years with overweight or obesity and isolated impaired fasting glucose. Intervention participants will adhere to an 8-week low-calorie dietary (LCD) regimen (~1,320 kcal/day) comprising specific macronutrient proportions (55% carbohydrate, 13% fat, 25% protein, and 2% fiber). Control participants will maintain their habitual dietary habits and physical activity levels. Primary outcomes at 8 weeks include between-group changes in weight, fasting plasma glucose, indices of ß-cell function and hepatic insulin resistance, and alanine aminotransferase levels. Secondary outcomes are feasibility metrics (response rate, screening yield, enrollment rate, intervention compliance, cost, staff time, and retention rate) and intervention acceptability. Qualitative research will explore facilitators, barriers, acceptability, satisfaction, and participant experiences with the LCD intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 35 to 65 years
2. Overweight (body mass index (BMI) ≥25 to <29 kg/m² or ≥23 to <29 kg/m² if Asian descent) or Obese (BMI ≥30 kg/m²)
3. Physically inactive (<150 minutes per week of moderate-intensity physical activity or <75 minutes per week of vigorous-intensity physical activity)
4. Prediabetes diagnosis or score ≥5 on the American Diabetes Association (ADA) risk tool

Exclusion Criteria:

1. Diagnosed with type 1 or type 2 diabetes
2. Cardiovascular disease (myocardial infarction, stroke, angina, heart failure, or other cardiac conditions)
3. Chronic kidney disease
4. Chronic liver disease (e.g., cirrhosis)
5. Cancers
6. Acute inflammatory bowel disease, irritable bowel syndrome, celiac disease, chronic pancreatitis, or other disorders potentially causing malabsorption
7. Food allergies
8. Participation in weight loss programs in the past six months
9. Currently following a specific diet (e.g., ketogenic diet, Mediterranean diet)
10. Participation in any exercise programs in the past six months
11. Currently taking weight-loss medications or drugs known to affect glycemia (steroids and antipsychotics)
12. Previous bariatric surgery or plan to have bariatric surgery during the study period
13. Planning to relocate during the study period
14. Intending to fast during the study period for religious or other reasons
15. Pregnancy or planning to become pregnant during the study period
16. Breastfeeding
17. Non-English speaker

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | Baseline
  Response rate is defined as the proportion of individuals responding to the invitation sent via the Epic database.
Screening yield | Baseline
  Screening yield: Proportion of screened individuals meeting eligibility criteria.
Enrollment rate | Baseline
  Enrollment rate: Proportion of eligible individuals who enroll in the study.
Resource utilization | Throughout the study period, an average of 10 weeks
  Resource utilization: Assessment of expenditures and staff time.
Retention rate | 4 and 8 weeks
  Retention rate: Proportion of enrolled participants who complete the study.
Intervention acceptability | 4 and 8 weeks
  Intervention acceptability will be assessed using the Theoretical Framework of Acceptability questionnaire. Scores range from 7 to 35. Higher scores indicate better acceptability among participants.
Feasibility of intervention | 4 and 8 weeks
  Will be assessed using the Feasibility of Intervention Measure questionnaire. Scores range from 4 to 20. Higher scores indicate better feasibility among participants.
Intervention appropriateness | 4 and 8 weeks
  Will be assessed with the Intervention Appropriateness Measure questionnaire. Scores range from 4 to 20. Higher scores indicate better appropriateness among participants.
Facilitators, barriers, acceptability, satisfaction, and participant experiences with the the intervention | 4 and 8 weeks
  Qualitative in-depth interviews

SECONDARY OUTCOMES:
Weight in kg | 4 and 8 weeks
  Weight will be measured using a digital weighing scale with an accuracy to the nearest 0.1 kg
Fasting plasma glucose in mg/dl | 4 and 8 weeks
  Will be analyzed by enzymatic assays
Indices of ß-cell function | 4 and 8 weeks
  Will be assessed using the insulinogenic index (IGI)
ß-cell function assessed by Oral Disposition Index (DI(O)) | 4 and 8 weeks
  Will be assessed using the Oral Disposition Index (DI(O))
ß-cell function assessed by Homeostatic Model Assessment of ß-cell Function (HOMA-B) | 4 and 8 weeks
  Will be assessed using the Homeostatic Model Assessment of ß-cell Function (HOMA-B)
Indices of hepatic insulin resistance | 4 and 8 weeks
  Will be assessed using the Hepatic Insulin Resistance Index (HIRI)
Alanine aminotransferase (liver enzyme) in U/L | 4 and 8 weeks
  Will be analyzed with colorimetric assays

CONTACTS AND LOCATIONS:
Overall Officials: Sathish Thirunavukkarasu, PhD, Principal Investigator — Emory University
Locations (1):
- Georgia Clinical & Translational Science Alliance (CTSA) Clinical Research Centers (GCRCs), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No